CLINICAL TRIAL: NCT00056537
Title: An Open-Label, Phase I, Repeat Dose-Escalation Study of ABR-217620 in Patients With Advanced Non-Small Cell Lung Cancer, Renal Clear Cell Carcinoma or Pancreatic Cancer
Brief Title: ABR-217620 in Patients With Advanced Non-Small Cell Lung Cancer, Renal Clear Cell Carcinoma or Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Active Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01762001
Record Dates: First submitted 2003-03-16; First posted 2003-03-18 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Non-Small-Cell Lung Carcinoma; Renal Cell Carcinoma; Pancreatic Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Pancreatic Neoplasms | interventions — naptumomab estafenatox; CD3 Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ABR-217620

INTERVENTIONS:
Drug: ABR-217620 — Starting dose: 0.5 mcg/kg; subsequent doses: individual, based on pre-treatment level of anti-SEA/E-120, body weight, and toxicities observed in prior patients on study; IV; one bolus injection each day for 5 consecutive days; up to 3 cycles
  Other Names: CD3; 5T4FabV18-SEA/E-120; naptumomab estafenatox; Anyara

SUMMARY:
The drug ABR-217620 is a combination of two proteins, one that recognizes tumor cells and one that triggers an attack on the tumor cells by activating some white blood cells belonging to the body's normal immune system. In animals, this results in an accumulation of white blood cells in the cancer that can fight the cancer. This study will test how much of the drug can be given to patients with non-small cell lung cancer, renal clear cell carcinoma, or pancreatic cancer without causing unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed non-small cell lung cancer, which is refractory to (progressed on or following) currently available standard therapies. Patients must have received (or declined) at least one standard regimen for advanced/metastatic disease.
* ECOG performance status of 0 or 1.
* Adequate bone marrow function as defined by absolute neutrophil count greater than or equal to 1500/mm3, and platelets greater than or equal to 100,000/mm3, and hemoglobin greater than or equal to 10 g/dL.
* Adequate renal function: creatinine less than or equal to 1.5 x upper limit of normal.
* Adequate hepatic function: bilirubin less than or equal to 2 x upper limit of normal, and SGOT (S-ASAT) and SGPT (S-ALAT) less than or equal to 2.5 x upper limit of normal.
* Life expectancy greater than 3 months.

Exclusion Criteria:

* Pregnant or breast-feeding women, or women of childbearing potential unless effective methods of contraception are used.
* A serious uncontrolled medical disorder or active infection that would impair the patient's ability to receive study treatment.
* History of or any concurrent malignancy, with the exception of the following malignancies, which may still be included: non-melanoma skin cancer, cervical cancer in situ, DCIS or LCIS of breast, past history of resected melanoma without clinical evidence of recurrent melanoma, past history of prostate cancer without clinical evidence of disease (includes patients receiving hormonal therapy).
* History of brain metastases, unless stable for more than 4 weeks, and not requiring steroid therapy and without clinical symptoms of brain metastases.
* Acute illness or evidence of infection, including unexplained fever (temperature greater than 100.5 degrees Fahrenheit or 38.1 degrees Celsius).
* Significant symptomatic cardiac disease including: history (within the past 6 months) or current unstable angina, congestive heart failure, or myocardial infarction; or patients with uncontrolled hypertension, or hypertension that is controlled only with multiply drugs (control by monotherapy is permitted).
* History of or current arrhythmias requiring treatment, with the exception of non-specific, asymptomatic ST-T wave changes or extrasystoles.
* History of cerebrovascular accident within the past 5 years.
* Seizure disorder requiring therapy.
* Treatment with beta-blockers, including topical therapy for glaucoma, during the 6-day treatment period (5 days' treatment + 1 day in patient follow-up), and within five days prior to start of treatment.
* Simultaneous participation in any other study involving investigational drugs or having participated in a study less than 4 weeks prior to start of study treatment.
* Treatment with systemic or inhaled corticosteroids within 2 weeks prior to the start of treatment.
* Treatment with anticoagulants, except when used to maintain the patency of a central venous line.
* Active autoimmune disease requiring therapy or any history of systemic lupus erythematosus or rheumatoid arthritis.
* Chemo/radio/immunotherapy less than 4 weeks (6 weeks for mitomycin C and nitrosoureas) before start of treatment.
* Major surgery less than 3 weeks.
* Known positive serology for HIV (patients with a known history of HIV will be excluded because of potential for unforeseen toxicity and morbidity in the immunocompromised host).
* Known chronic Hepatitis B or C.
* Previous exposure to murine monoclonal antibody (with HAMA titer above detection limit at baseline) or known hypersensitivity to murine proteins.
* Patients currently on renal dialysis treatment.
* Known allergy or hypersensitivity to aminoglycosides e.g. kanamycin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) as a function of pre-treatment anti-SEA/E-120 levels | 56 days after start of first treatment cycle

SECONDARY OUTCOMES:
Safety profile | During or after first treatment cycle, second treatment cycle, later cycles if available
Pharmacokinetic parameters | Days 1 and 5 of each cycle
Immunological response | Days 28 and 56 of first and second treatment cycles, later cycles if available
Objective response rate | Days 28 and 56 of first and second treatment cycles, later cycles if available
Time to progression and Survival | Followed for up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Kilany, Study Director — Active Biotech AB
Locations (3):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States
- Det Norske Radiumhospitalet, Oslo, Norway
- Paterson Institute for Cancer Research, Christie Hospital NHS Trust and Research Institute, Manchester, United Kingdom